CLINICAL TRIAL: NCT05081544
Title: Impact of Multi-tasking Situations on the Dismounted Soldier's Cognitive Load
Acronym: SiMuCCoDé
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PBMD01; 2021-A00733-38 (Other: IDRCB)
Record Dates: First submitted 2021-10-07; First posted 2021-10-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Load
Keywords: cognitive load

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increased complexity of the dismounted combatant's equipment can result in a strain on the various senses (e.g., visual, auditory) that can exceed an individual's limited information processing abilities. The combatant may thus be cognitively overloaded in multi-tasking operational situations.

There has been a great deal of research conducted on cognitive load. A battery of multitasking tests has been developed in the field of aeronautics, but, to our knowledge, no measurement of cognitive load specifically dedicated to combatants has been conducted yet.

ELIGIBILITY:
Inclusion Criteria:

* be a group leader in an infantry regiment,
* be over 18 years old.

Exclusion Criteria:

* be a woman,
* have a heart condition,
* have a visual disease not corrected by glasses or contact lenses,
* have a hearing score ≥ 2 on the SIGYCOP,
* have a psychiatric disorder, a progressive neurological or organic disease requiring drug treatment,
* take psychotropic drugs,
* take more than 28 units of alcohol per week.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of healthy volunteers from several French infantry regiments (group leaders).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive load level | At enrollment (Day 1)
  Cognitive load level will be measured using NASA-TLX questionnaire. NASA-TLX questionnaire comprises 6 dimensions (mental demands, physical demands, time demands, performance, effort and frustration). Each dimension has a score ranging from 0 (low cognitive load) to 100 (high cognitive load), except for the "performance" dimension, whose score ranges from 0 (good performance) to 100 (low performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided